CLINICAL TRIAL: NCT02007785
Title: Determining the Applicability of the Cognitive Orientation to Daily Occupational Performance (CO-OP) as a Meta-Cognitive Rehabilitation Strategy for Individuals With Parkinson's Disease-Related Cognitive Impairment
Brief Title: Study of the Effect of the Cognitive Orientation to Daily Occupational Performance (CO-OP) on Cognitive Impairment in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Catherine Bryden Dueck, O.T. Reg. (MB), graduate student, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2013:400
Record Dates: First submitted 2013-11-14; First posted 2013-12-11 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Parkinson's Disease; Cognitive Impairment
Keywords: Cognitive Orientation to daily Occupational Performance; CO-OP
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

ARMS (1):
- CO-OP treatment protocol (Experimental): Participants with Parkinson's disease will be participating in up to 12 one-on-one treatment sessions with 2 sessions per week, for up to 6 weeks. Each session will last 45-60 minutes. During these treatment sessions, each participant will be taught a problem-solving strategy that teaches individuals to monitor and adjust their own actions. Participants will be guided by the principal investigator to select 5 individual treatment goals to work on during treatment. Sessions will continue until all 5 treatment goals have been met or until 12 sessions have been completed, whichever occurs earlier. Initially, each participant's respective primary caregiver will be required to attend treatment sessions, so that the caregiver may be familiar with the treatment strategy in order to coach the participant with Parkinson's disease when you he or she uses the strategy at home.
  Interventions: Behavioral: CO-OP treatment protocol

INTERVENTIONS:
Behavioral: CO-OP treatment protocol — Participants with Parkinson's disease will be participating in up to 12 one-on-one treatment sessions with 2 sessions per week, for up to 6 weeks. Each session will last 45-60 minutes. During these treatment sessions, each participant will be taught a problem-solving strategy that teaches individuals to monitor and adjust their own actions. Participants will be guided by the principal investigator to select 5 individual treatment goals to work on during treatment. Sessions will continue until all 5 treatment goals have been met or until 12 sessions have been completed, whichever occurs earlier. Initially, each participant's respective primary caregiver will be required to attend treatment sessions, so that the caregiver may be familiar with the treatment strategy in order to coach the participant with Parkinson's disease when you he or she uses the strategy at home.
  Other Names: Cognitive Orientation to daily Occupational Performance

SUMMARY:
The purpose of the study will be to determine the effects of the Cognitive Orientation to daily Occupational Performance (CO-OP) as a treatment program for individuals with Parkinson's disease-related cognitive impairment. The potential effects of the CO-OP on successful engagement in meaningful activities will be examined from participants' and live-in caregivers' perspectives. Effects of the CO-OP on participant-perceived health-related quality of life and caregiver burden will also be evaluated.

Hypotheses:

1. Training with the CO-OP will have an effect or multiple effects on participation in meaningful activities and health-related quality of life for individuals with Parkinson's-related cognitive impairment.
2. Training with the CO-OP will have an effect or multiple effects on caregiver burden and health-related quality of life for caregivers of individuals with Parkinson's-related cognitive impairment.

ELIGIBILITY:
Inclusion Criteria for Participants with Parkinson's disease:

* Clinical diagnosis of Idiopathic Parkinson's Disease
* Presence of a live-in caregiver or significant other who is willing to participate in the study
* Montreal Cognitive Assessment (MoCA) score above 16/30 and below 26/30
* Schwab and England Activities of Daily Living Scale scores between 60% and 90%
* Hoehn and Yahr Scale scores between Stage 1 and Stage 3
* Self-reported difficulty completing routine functional activities that may be related to new cognitive changes since PD diagnosis

Exclusion Criteria for Participants with Parkinson's disease:

* Clinical diagnosis of atypical parkinsonism
* Clinical diagnosis of young-onset Parkinson's disease
* Co-morbidities associated with cognitive impairment
* Poorly controlled depression
* Clinical diagnosis of dementia
* Residence outside boundaries of the city of Winnipeg, Manitoba, Canada

Inclusion Criteria for Caregiver Participants:

* Live in the same residence as participant with Parkinson's
* Be willing to participate

Exclusion Criteria for Caregiver Participants:

* Scores at or below 16/30 on Montreal Cognitive Assessment (MoCA)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change from Pre-Intervention Phase Baseline Pattern (2 week duration) on Canadian Occupational Performance Measure (COPM) score pattern at Intervention Phase (6 week duration), Post-Intervention Phase (2 week duration), and 3-Month Follow-up | Pre-Intervention Phase: Days 1, 3, 5, 9 and 11; Intervention Phase: Following treatment sessions 2, 4, 6, 8, and 10; Post-Intervention Phase: Days 1, 3, 5, 9, and 11; Follow-Up Phase: 3 months after completion of Post-Intervention Phase
  The COPM is a semi-structured interview focusing on client-centred problem identification that is founded on the Canadian guidelines for client-centred occupational therapy practice and requires approximately 30-40 minutes to administer. The COPM consists of three sections: self-care (basic and instrumental activities of daily living); productivity (education and work); and leisure (play, leisure, and social participation). The assessment begins with self-report of occupational performance issues. The identified occupational performance issues are then rated by the client according to importance on a 10-point Likert scale. The five issues identified as most important to the client are then rated again according to the client's self-determined performance level and satisfaction. Since the COPM is designed to be used as a measure of change, performance and satisfaction levels are scored again after a period of time, (usually during which an intervention has been administered).
Change from Pre-Intervention Phase Baseline Pattern (2 week duration) on Parkinson Disease Questionnaire - 39 (PDQ-39) score pattern at Intervention Phase (6 week duration), Post-Intervention Phase (2 week duration), and 3-Month Follow-Up | Pre-Intervention Phase: Days 1, 3, 5, 9, and 11; Intervention Phase: Following treatment sessions 2, 4, 6, 8, and 10; Post-Intervention Phase: Days 1, 3, 5, 9, and 11; Follow-Up Phase: 3 months after completion of Post-Intervention Phase
  The PDQ-39 is the most widely used Parkinson's-specific measure of health-related quality of life. It is a self-administered questionnaire containing thirty nine questions that cover eight aspects of health-related quality of life: mobility (10 items), activities of daily living (6 items), emotional well-being (6 items), stigma (4 items), social support (3 items), cognition (4 items), communication (3 items), and bodily discomfort (3 items). Patients are asked to select the frequency of each problem item occurring over the past month on a 5-point scale (never / occasionally / sometimes / often / always or cannot do at all). The PDQ-39 requires approximately 10-20 minutes to administer.
Change from Pre-Intervention Phase Baseline Pattern (2 week duration) on Zarit Burden Interview score pattern at Intervention Phase (6 week duration), Post-Intervention Phase (2 week duration), and 3-Month Follow-Up | Pre-Intervention Phase: Days 1, 3, 5, 9, and 11; Intervention Phase: Following treatment sessions 2, 4, 6, 8, and 10; Post-Intervention Phase: Days 1, 3, 5, 9, and 11; Follow-Up Phase: 3 months after completion of Post-Intervention Phase
  The Zarit Burden Interview (ZBI) is the most widely used measure of caregiver burden. It is a self-administered 22-item questionnaire designed to assess caregivers' perceptions of burden related to caring for an older person with dementia or a person with a disability. Questions on the interview address caregivers' physical health, as well as emotional, social, and financial wellbeing. Caregivers are asked to select the frequency of each problem item on a 5-point scale (never / rarely / sometimes / quite frequently / nearly always). The ZBI takes approximately 5-10 minutes to administer.
Change from Pre-Intervention Baseline Observations (2 week duration) on Direct Observation Record at Intervention Phase (6 week duration), Post-Intervention Phase (2 week duration), and 3-Month Follow-Up | Pre-Intervention Phase: Day 1; Intervention Phase: during all treatment sessions (1-12) as well as during an interview session between treatment sessions 6 and 7; Post-Intervention Phase: Day 1; Follow-Up Phase: Day 1
  Field notes consisting of direct observations of the behaviours of study participants and their caregivers / significant others and relevant contextual events and environmental features will be recorded with detailed descriptions in a log book. Observational data collected during the proposed study will provide rich,detailed information related to interactions between study participants and the physical and social environments in which the participants will work toward their CO-OP treatment goals, as well as detailed information related to the participants' performance on self-selected CO-OP treatment goals. Examples of observations that will be recorded include non-verbal body language, facial expression, and tone of voice of participants and caregivers, and detailed descriptions of physical environmental aspects that are relevant to the context of the study session.
Change from Pre-Intervention Baseline Observations (2 week duration) on Semi-Structured Interview at Intervention Phase (6 week duration), Post-Intervention Phase (2 week duration), and 3-Month Follow-Up | Pre-Intervention Phase: Day 1; Intervention Phase: between treatment sessions 6 and 7; Post-Intervention Phase: Day 1; Follow-Up Phase: Day 1
  Semi-structured interviews will resemble guided conversations using an interview guide consisting of open-ended questions. When appropriate, the interviewer will ask value neutral probing follow-up questions in order to elicit more information from the interviewee. Appropriate situations in which probing follow-up questions may be asked include when examples, explanations, and rationales for interviewees' responses are necessary to capture the participants' beliefs and views as thoroughly and accurately as possible. The interviewees' verbal statements will be recorded verbatim in an interview log book. Observations regarding body language and affect will also be recorded in the log book. Interviews will be audio recorded using two digital recorders (in case of failure of one recorder) in order to have as much data as possible available for analysis and to verify the accuracy of the data collected.
Reflective Journal Log | From Day 1 of Baseline Phase until completion of Follow-Up Phase (up to 26 weeks in total)
  A reflective journal log will be maintained as a deliberate, systematic self-examination process for the principal investigator. The principal investigator's thoughts, feelings, and reactions related to questions, quandaries, and complexities that arise as the study progresses will be recorded. Awareness of this data is important to identify and account for its potential to bias the processes of data collection and analysis, which may also influence emerging interpretations of study results.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine E Bryden Dueck, BMR (OT), Principal Investigator — University of Manitoba
Locations (1):
- Deer Lodge Centre, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Calleo J, Burrows C, Levin H, Marsh L, Lai E, York MK. Cognitive rehabilitation for executive dysfunction in Parkinson's disease: application and current directions. Parkinsons Dis. 2012;2012:512892. doi: 10.1155/2012/512892. Epub 2011 Nov 2. PMID 22135762
- [Background] Dawson DR, Gaya A, Hunt A, Levine B, Lemsky C, Polatajko HJ. Using the cognitive orientation to occupational performance (CO-OP) with adults with executive dysfunction following traumatic brain injury. Can J Occup Ther. 2009 Apr;76(2):115-27. doi: 10.1177/000841740907600209. PMID 19456090
- [Background] DePoy, E., & Gitlin, L. (2005). Case Study Designs. In E. DePoy, & L. Gitlin, Introduction to Reserach: Understanding and Applying Multiple Strategies (3rd Ed.) (pp. 277-283). St. Louis, MO: Mosby.
- [Background] Disbrow EA, Russo KA, Higginson CI, Yund EW, Ventura MI, Zhang L, Malhado-Chang N, Woods DL, Sigvardt KA. Efficacy of tailored computer-based neurorehabilitation for improvement of movement initiation in Parkinson's disease. Brain Res. 2012 May 3;1452:151-64. doi: 10.1016/j.brainres.2012.02.073. Epub 2012 Mar 9. PMID 22459048
- [Background] Emre M, Aarsland D, Brown R, Burn DJ, Duyckaerts C, Mizuno Y, Broe GA, Cummings J, Dickson DW, Gauthier S, Goldman J, Goetz C, Korczyn A, Lees A, Levy R, Litvan I, McKeith I, Olanow W, Poewe W, Quinn N, Sampaio C, Tolosa E, Dubois B. Clinical diagnostic criteria for dementia associated with Parkinson's disease. Mov Disord. 2007 Sep 15;22(12):1689-707; quiz 1837. doi: 10.1002/mds.21507. PMID 17542011
- [Background] Foster ER, Hershey T. Everyday Executive Function Is Associated With Activity Participation in Parkinson Disease Without Dementia. OTJR (Thorofare N J). 2011;31(1):16-22. doi: 10.3928/15394492-20101108-04. PMID 21921994
- [Background] Hoops S, Nazem S, Siderowf AD, Duda JE, Xie SX, Stern MB, Weintraub D. Validity of the MoCA and MMSE in the detection of MCI and dementia in Parkinson disease. Neurology. 2009 Nov 24;73(21):1738-45. doi: 10.1212/WNL.0b013e3181c34b47. PMID 19933974
- [Background] Leroi I, Collins D, Marsh L. Non-dopaminergic treatment of cognitive impairment and dementia in Parkinson's disease: a review. J Neurol Sci. 2006 Oct 25;248(1-2):104-14. doi: 10.1016/j.jns.2006.05.021. Epub 2006 Jun 27. PMID 16806271
- [Background] Mohlman J, Chazin D, Georgescu B. Feasibility and acceptance of a nonpharmacological cognitive remediation intervention for patients with Parkinson disease. J Geriatr Psychiatry Neurol. 2011 Jun;24(2):91-7. doi: 10.1177/0891988711402350. PMID 21546649
- [Background] Paris AP, Saleta HG, de la Cruz Crespo Maraver M, Silvestre E, Freixa MG, Torrellas CP, Pont SA, Nadal MF, Garcia SA, Bartolome MV, Fernandez VL, Bayes AR. Blind randomized controlled study of the efficacy of cognitive training in Parkinson's disease. Mov Disord. 2011 Jun;26(7):1251-8. doi: 10.1002/mds.23688. Epub 2011 Mar 25. PMID 21442659
- [Background] Polatajko, H., & Mandich, A. (2004). Enabling Occupation in Children: The Cognitive Orientation to daily Occupational Performance (CO-OP) Approach. Ottawa: CAOT Publications ACE.
- [Background] Sammer G, Reuter I, Hullmann K, Kaps M, Vaitl D. Training of executive functions in Parkinson's disease. J Neurol Sci. 2006 Oct 25;248(1-2):115-9. doi: 10.1016/j.jns.2006.05.028. Epub 2006 Jun 12. PMID 16765378
- [Background] Sinforiani E, Banchieri L, Zucchella C, Pacchetti C, Sandrini G. Cognitive rehabilitation in Parkinson's disease. Arch Gerontol Geriatr Suppl. 2004;(9):387-91. doi: 10.1016/j.archger.2004.04.049. PMID 15207437
- [Background] Skidmore ER, Holm MB, Whyte EM, Dew MA, Dawson D, Becker JT. The feasibility of meta-cognitive strategy training in acute inpatient stroke rehabilitation: case report. Neuropsychol Rehabil. 2011 Apr;21(2):208-23. doi: 10.1080/09602011.2011.552559. PMID 21391121
- [Background] Vale S. Current management of the cognitive dysfunction in Parkinson's disease: how far have we come? Exp Biol Med (Maywood). 2008 Aug;233(8):941-51. doi: 10.3181/0707-MR-193. Epub 2008 Jun 5. PMID 18535172